CLINICAL TRIAL: NCT03188705
Title: Enrichment of CES1 Carriers in the Pharmacogenomics Anti-Platelet Intervention Study
Brief Title: CES1 Carriers in the PAPI Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Joshua Lewis, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00075567
Record Dates: First submitted 2017-06-14; First posted 2017-06-15 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Heart Diseases; Coronary Disease; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia; Artery Occlusion; Aspirin Sensitivity; Clopidogrel, Poor Metabolism of; Platelet Dysfunction; Platelet Thrombus
Keywords: pharmacogenetics; carboxylesterase; Personalized Medicine
MeSH Terms: conditions — Heart Diseases; Coronary Disease; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia; Arterial Occlusive Diseases | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: The investigators will enroll up to 50 healthy Amish participants who have been identified through existing whole genome and exome sequencing along with bioinformatic approaches that have genetic variants that are predicted to significantly impact CES1 expression or catalytic function. Enrolled participants will undergo a two-stage intervention with clopidogrel (300 mg loading dose then 75 mg per day for the next 6 days), followed by clopidogrel (75 mg) plus aspirin 324 mg for 1 day. Platelet aggregation studies and other measures of platelet function will be performed before and after each intervention. In combination with previously collected data as part of the PAPI Study, the investigators will then characterize the impact of genetic variation in CES1 on clopidogrel and dual antiplatelet therapy response through single- and multi-variant association modeling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Overall Cohort (Experimental): Participants will receive clopidogrel treatment alone (300 mg loading dose followed by 75 mg/d for 6 days), followed by clopidogrel (75 mg) plus aspirin (324 mg) treatment on day 8.
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Participants will receive 300 mg of clopidogrel on the first day, then 75 mg per day for the next 6 days. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Other Names: Plavix
Drug: Aspirin — Participants will receive a single dose of 324 mg aspirin on the last day of clopidogrel administration.

SUMMARY:
This study builds, in part, upon preliminary results generated as part of the Pharmacogenomics Anti-Platelet Intervention (PAPI) Study (NCT00799396). The purpose of this investigation is to assess the impact of genetic variation in the carboxylesterase 1 (CES1) on response to clopidogrel as well as dual antiplatelet therapy (i.e. clopidogrel and aspirin), as assessed by ex vivo platelet aggregometry, in healthy Amish individuals. The investigators hypothesize that participants who carry alleles that modify the activity or expression of CES1 will have altered response to clopidogrel as well as dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* Of Old Order Amish descent

Exclusion Criteria:

* Currently pregnant or less than 6 months have passed since delivery
* Currently breast feeding
* Has a history of a bleeding disorder or major spontaneous bleed, such as peptic ulcer, epistasis, or intracranial bleed
* Has severe hypertension, defined by a blood pressure above 160/95 mm Hg
* Takes medications that would affect the outcome(s) to be measured and cannot willingly and safely, in the opinion of the treating physician and study physician, discontinue these medications for 1 week prior to protocol initiation
* Is taking vitamins or other supplements and is unwilling to discontinue use for at least 1 week prior to study
* Has a coexisting malignancy
* Has a creatinine level greater than 2.0 mg/dl, aspartate transaminase (AST) or alanine transaminase (ALT) greater than two times the upper limit of normal, hematocrit less than 32%, or a thyroid-stimulating hormone (TSH) less than 0.4 or greater than 5.5 mIU/L
* Has a bleeding disorder or history of gastrointestinal bleeding or other major bleeding episode
* Is currently taking aspirin, clopidogrel, or anti-coagulants, such as warfarin, heparin, or GPIIb/IIIa antagonists, and have conditions that might place the participant at increased risk from withdrawal of these medications 14 days prior to protocol initiation
* History of unstable angina, heart attack, angioplasty (including stent placement), coronary artery bypass surgery, atrial fibrillation, stroke or transient ischemic attacks, diabetes, or deep vein thrombosis or other thrombosis
* Has polycythemia, or thrombocytosis, defined by a platelet count greater than 500,000
* Has thrombocytopenia, defined by a platelet count less than 75,000
* Has had surgery within the last 6 months
* Has an aspirin or clopidogrel allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Lewis, PhD, Principal Investigator — University of Maryland
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes
  It is possible that deidentified data will be deposited into large public databases as per NIH data sharing policies (e.g. dbGAP, PharmGKB). Data to be shared would include, but not limited to, anthropometric data, study outcome data, and relevant covariate data used in statistical models of association. It is anticipated that data would be available after the completion of the trial. The data will be obtained from the participants and the study-related research procedures.

RESULTS

PARTICIPANT FLOW:
Groups:
- Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment: Participants will receive clopidogrel treatment alone (300 mg loading dose followed by 75 mg/d for 6 days), followed by clopidogrel (75 mg) plus aspirin (324 mg) treatment on day 8.
  Clopidogrel: Participants will receive 300 mg of clopidogrel on the first day, then 75 mg per day for the next 6 days. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Aspirin: Participants will receive a single dose of 324 mg aspirin on the last day of clopidogrel administration.
Period: Clopidogrel Treatment
Arm/Group | Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Clopidogrel Plus Aspirin Treatment
Arm/Group | Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Platelet Function in Response to Clopidogrel
Description: Baseline minus post clopidogrel/pre-aspirin platelet rich plasma (PRP) maximum aggregation in response to ADP (20 ug/ml) or collagen (5 ug/ml). Maximum platelet aggregation is recorded by the platelet aggregometer as a percentage. Data shown below represent the maximum platelet aggregation value obtained at baseline (recorded as a percentage) minus the maximum platelet aggregation value obtained after clopidogrel administration but before aspirin administration (also recorded as percentage). Thus, values recorded below represent a percentage change.
Time Frame: Measured at baseline and after 8 days of clopidogrel treatment
Measure: Mean (Standard Deviation); unit: percentage of maximum aggregation change
Arm/Group | Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment
Number analyzed (Participants) | 5
percentage of maximum aggregation change
  Change in the percentage of maximal platelet aggregation in response to 20 ug/ml ADP | 37.4 (5.5)
  Change in the percentage of maximal platelet aggregation in response to 5 ug/ml collagen | 20.4 (7.9)

2. Primary Outcome: Changes in Platelet Function in Response to Clopidogrel Plus Aspirin
Description: Baseline minus post clopidogrel/post-aspirin platelet rich plasma (PRP) maximum aggregation in response to ADP (20 ug/ml) or collagen (5 ug/ml). Maximum platelet aggregation is recorded by the platelet aggregometer as a percentage. Data shown below represent the maximum platelet aggregation value obtained at baseline (recorded as a percentage) minus the maximum platelet aggregation value obtained after clopidogrel and aspirin administration (also recorded as percentage). Thus, values recorded below represent a percentage change.
Time Frame: Measured at baseline and after 8 days clopidogrel administration plus 1 day of aspirin treatment
Measure: Mean (Standard Deviation); unit: percentage of max aggregation change
Arm/Group | Clopidogrel Alone Followed by Clopidogrel and Aspirin Treatment
Number analyzed (Participants) | 5
percentage of max aggregation change
  Change in the percentage of maximal platelet aggregation in response to 20 ug/ml ADP | 38.0 (8.2)
  Change in the percentage of maximal platelet aggregation in response to 5 ug/ml collagen | 55.8 (8.8)

ADVERSE EVENTS:
Time Frame: 37 days
Description: Adverse event data were collected during both intervention periods and for 30 days after the final study visit.
Groups:
- Clopidogrel Alone Treatment; Clopidogrel and Aspirin Treatment: All participants will receive clopidogrel treatment alone (300 mg loading dose followed by 75 mg/d for 6 days), followed by clopidogrel (75 mg) plus aspirin (324 mg) treatment on day 8.
  Clopidogrel: Participants will receive 300 mg of clopidogrel on the first day, then 75 mg per day for the next 6 days. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Aspirin: Participants will receive a single dose of 324 mg aspirin on the last day of clopidogrel administration.
Arm/Group | Clopidogrel Alone Treatment | Clopidogrel and Aspirin Treatment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03188705/Prot_SAP_000.pdf